CLINICAL TRIAL: NCT00007267
Title: Psychosocial Interventions for Scleroderma
Brief Title: Psychological Treatments for Scleroderma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR047219 (NIH); R01AR047219 (NIH); NIAMS-056
Record Dates: First submitted 2000-12-16; First posted 2000-12-18 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Pain; Depression; Scleroderma; Systemic Sclerosis
Keywords: Scleroderma; Systemic sclerosis; Depression; Pain; Disfigurement; Body image dissatisfaction; Cognitive-behavioral therapy; Self-help; Psychological intervention
MeSH Terms: conditions — Pain; Depression; Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive individual cognitive behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy
- 2 (Experimental): Participants will receive self-help cognitive behavioral intervention facilitated by a psychologist
  Interventions: Behavioral: Self-help cognitive behavioral intervention facilitated by a psychologist
- 3 (Active Comparator): Participants will receive a disease/health education intervention
  Interventions: Behavioral: Disease/health education

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy
  Arms: 1
Behavioral: Disease/health education
  Arms: 3
Behavioral: Self-help cognitive behavioral intervention facilitated by a psychologist
  Arms: 2

SUMMARY:
This study will examine the effectiveness of two psychological treatment approaches designed to help people who have scleroderma with three important areas of daily living: pain, depression, and distress about changes in appearance. The study will also evaluate the impact of depression on the two psychological treatments. Because psychological approaches requiring a trained professional can be expensive and are often not available to most patients, this study will also look at the effectiveness of a self-help treatment approach.

DETAILED DESCRIPTION:
This study will examine the efficacy of psychological interventions designed to target important areas of daily living for people with scleroderma: pain, depression, and distress about disfigurement. The study will also examine the effect of clinical depression on impact of the psychological treatments. Because psychological interventions requiring a trained professional can be costly and are often not available to the majority of patients, the study will also examine the efficacy of a self-help intervention.

The study will recruit 201 patients with systemic sclerosis who report symptoms of pain, depression, or distress about disfigurement and will randomly assign them to one of three interventions: individual cognitive behavioral therapy, self-help cognitive behavioral intervention facilitated by a psychologist, or a disease/health education intervention. An individual blinded to intervention assignment will collect measures of pain, functioning, distress about disfigurement, and mood at baseline and following the 8-week intervention period.

Both the cognitive-behavioral self-help materials and the educational materials (eight written chapters and audiotapes) will be designed for home use but will be supplemented by two individual sessions and two telephone contacts with the professional. Patients will be followed for 1 year after completing the active intervention phase.

These findings will increase understanding of the quality of life of individuals with scleroderma and determine whether self-help interventions can be used effectively to manage pain, depression, and distress about disfigurement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CREST or systemic sclerosis
* Short-Form McGill Pain Questionnaire score 6 or higher
* Satisfaction with Appearance score of 15 or higher
* Beck Depression score of 10 or higher

Exclusion Criteria:

* Patients reporting severe depression with suicidal ideation
* Delirium, dementia, or cognitive impairment (Mini Mental State Examination (MMSE) < 24))
* Terminal illness with a life expectancy of less than 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2001-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Measured at Week 8

SECONDARY OUTCOMES:
Body image dissatisfaction | Measured at Week 8
Pain | Measured at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Haythornthwaite, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Haythornthwaite JA, Heinberg LJ, McGuire L. Psychologic factors in scleroderma. Rheum Dis Clin North Am. 2003 May;29(2):427-39. doi: 10.1016/s0889-857x(03)00020-6. PMID 12841303